CLINICAL TRIAL: NCT04671706
Title: Effectiveness, Tolerability, and Safety of Belimumab in Patients With Systemic Lupus Erythematosus Treated at the Spanish Departments of Internal Medicine
Brief Title: Belimumab in Patients With Systemic Lupus Erythematosus
Acronym: BeliLES
Status: Not yet recruiting | Type: Observational
Sponsor: Grupo de Trabajo de Enfermedades Autoinmunes Sistémicas (GEAS) de la Fundación Española de Medicina (Other)
Responsible Party: Sponsor
Other Study IDs: BeliLES
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus; SLE; Belimumab
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The BeliLES-GEAS project pretends to obtain an extensive data registry of patients with systemic lupus erythematosus (SLE).

The main objective is to create a national SLE patients registry treated with belimumab to describe effectiveness and safety of intravenous (IV) or subcutaneous (SC) belimumab in patients with active SLE treated in the Spanish departments of Internal Medicine in a real-life setting. This research project aspires to cover the vast majority (if not the whole) of SLE patients treated with belimumab in all of the Spanish Departments of Internal Medicine.

DETAILED DESCRIPTION:
The goal of BeliLES-GEAS registry is to create an observational, non-randomized, non-controlled, national multicenter prospective and retrospective cohort with the aim to explore the real performance, with its lights and shadows, of Belimumab, either IV or SC, in a real-world population of lupus patients.

The intention is to perform a longer-term follow up, so that the measure of hard outcomes, such as improvement in mortality, could be feasible, but also reliable data regarding the safety profile could be recorded.

In order to achieve that, the following variables will be included: individual criteria as part of 2019 EULAR/ACR, SLICC or ACR 1997 classification criteria, gender, age at diagnosis, age at symptoms onset, duration of the disease, age at first Belimumab administration, mean time of follow-up prior to, and from Belimumab administration, complete medical history including other systemic autoimmune diseases, type/s of organ/systems affected by SLE, prior immunosuppressants received, number of flares 2 years prior Belimumab onset, number of medical visits, number of days of sick leave, type of disease, treatment and laboratory data. As a measure of damage, Systemic Lupus International Collaborating Clinics-Damage Index (SLICC-DI) score will be calculated at baseline and at 12, 18, 24 months and yearly of follow-up. All centers will be requested to provide the SLICC-DI calculated annually of the last five years before the initiation of belimumab, when available.

The efficacy will be evaluated as time to reach any of the definition of remission included in the DORIS (definitions of remission in SLE) consensus, or LLDAs (lupus low disease activity state). Regarding the safety of Belimumab in real-world setting, it will be defined and evaluated by documenting adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfillment of the 2019 EULAR/ACR classification criteria for SLE, SLICC classification criteria, 1997 American College of Rheumatology (ACR) revised criteria for SLE or patients with only 3 criteria but SLE diagnosed according to the clinical judgment of the treating physician.
2. Age of 18 years or more.
3. Having received at least one dose of intravenous or subcutaneous belimumab according the physician criteria regardless the clinical/immunological response.
4. Signed informed consent.

Exclusion Criteria:

1) Negative from the patient to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Systemic Lupus Erythematosus
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Disease activity, clinical outcomes, and describe overall patterns of SLE care | 2 years
  Study endpoints are clinically recognized (and objectively confirmed). Additional endpoints will be the identification of predictors of response in our patients

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Espinosa, Study Chair — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No